CLINICAL TRIAL: NCT06761287
Title: Role of Local Endoscopic Excision After Neoadjuvant Therapy in Locally Advanced Rectal Cancer: A Prospective Study
Brief Title: Optimizing Patient Selection for Surgery Using Pathologic Analysis Following Neoadjuvant Therapy in Locally Advanced Rectal Cancer
Acronym: OPAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Mariana Figueiredo, Medical Doctor (Gastroenterology, Therapeutic Endoscopy and Digestive Oncology), Centre Hospitalier Universitaire Saint Pierre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPAL202412
Record Dates: First submitted 2024-12-20; First posted 2025-01-07 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Locally Advanced Rectal Cancer (LARC)
Keywords: locally advanced rectal cancer; neoadjuvant; endoscopic resection; endoscopic submucosal dissection; endoscopic intermuscular dissection; feasibility; safety
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Complete clinical response (Experimental): Defined as the presence of residual clear scar seen on endoscopic examination, without evidence of invasive disease (>T2) or locoregional invasion on magnetic resonance imaging and without any signs of metastatic disease on a computerized tomography scan.
  Interventions: Procedure: Endoscopic resection
- Near complete clinical response (Experimental): Defined as the presence of irregular mucosa or small mucosal nodules or superficial ulceration or persisting erythema of the scar seen on endoscopic examination, without evidence of invasive disease (>T2) or locoregional invasion on magnetic resonance imaging and without any signs of metastatic disease on a computerized tomography scan.
  Interventions: Procedure: Endoscopic resection; Behavioral: Short interval restaging; Procedure: Total mesorectal excision
- Incomplete response with presence of superficial residual tissue (Experimental): Defined as the presence of superficial residual tissue without features of deep invasion seen on endoscopic examination, without evidence of invasive disease (>T2) or locoregional invasion on magnetic resonance imaging and without any signs of metastatic disease on a computerized tomography scan.
  Interventions: Procedure: Endoscopic resection; Behavioral: Short interval restaging; Procedure: Total mesorectal excision
- No significant response (Active Comparator): Persistant local signs of malignancy
  Interventions: Procedure: Total mesorectal excision

INTERVENTIONS:
Procedure: Endoscopic resection — Eligible patients will undergo endoscopic submucosal dissection (ESD) or endoscopic intermuscular dissection (EID) after two to eight weeks of nCRT completion, depending on the used neo-adjuvant regimen. Procedures will be performed using the GIF EZ-1500 endoscope (Olympus America, Center Valley, PA, USA) and an electrosurgical unit (VIO 300 D; Erbe, Germany) to power the electrosurgical knife (1.5-mm DualKnife J, Olympus America). For mucosal incision, Endocut or Drycut mode will be used, while Precise, Swift or Spray Coagulation modes will support submucosal dissection and hemostasis. An initial submucosal lift will be created by Glycéol Gel injection. The ERBE Flushing Pump (Erbe, Germany) will supply further submucosal lift during dissection through foot pedal-controlled, pressurized injections of methylene blue and saline solution delivered via the DualKnife J's ceramic-tipped tubing.
  Arms: Complete clinical response; Incomplete response with presence of superficial residual tissue; Near complete clinical response
Behavioral: Short interval restaging — Close follow-up and endoscopic re-evaluation four to eight weeks after the initial evaluation*.
  *Defined as the first endoscopic evaluation after completion of the neoadjuvant treatment
  Arms: Incomplete response with presence of superficial residual tissue; Near complete clinical response
Procedure: Total mesorectal excision — This technique consists of the surgical complete removal of the rectum, together with the surrounding mesorectum lymphovascular fatty tissue (mesorectum).
  Arms: Incomplete response with presence of superficial residual tissue; Near complete clinical response; No significant response

SUMMARY:
This interventional, non-randomized, prospective trial aims to evaluate the role of endoscopic resection following neoadjuvant treatment in patients with locally advanced rectal cancer.

Phase I focuses on assessing the feasibility, safety and efficacy of endoscopic resection of residual scar or superficial residual neoplastic tissue following neoadjuvant treatment.

Phase II explores the potential of this approach to guide patient selection for total mesorectal excision and to serve as a definitive treatment option for those with limited residual disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Signed informed consent
* Patients diagnosed with locally advanced rectal cancer showing complete or near-complete clinical response after neoadjuvant therapy without evidence of invasive disease (>T2) or locoregional invasion on magnetic resonance imaging and without any signs of metastatic disease on a computerized tomography scan.
* Patients diagnosed with locally advanced rectal cancer showing incomplete response with presence of superficial residual lesions, without invasive features on endoscopic evaluation, without evidence of invasive disease (>T2) or locoregional invasion on magnetic resonance imaging and without any signs of metastatic disease on a computerized tomography scan.
* Without previous medical history of rectal cancer or rectal surgery

Exclusion Criteria:

* Previous medical history of rectal cancer
* Previous rectal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Endoscopic Resection | From the endoscopic procedure date to the date of reported pathology results, estimated to a maximum of 15 days
  Feasibility of the endoscopic resection technique in the context of locally advanced rectal cancer treated with neoadjuvant therapy including radio-chemotherapy. This will be assessed by the curative, en-bloc, and R0 resection rates.
Disease Recurrence | From the endoscopic procedure date until 5 years after the completion of the neoadjuvant therapy
  This will be assessed by the rate of local or distant recurrences and the need of salvage surgery within 1, 3 and 5 years following the neoadjuvant treatment and endoscopic resection.

SECONDARY OUTCOMES:
Complete endoscopic resection rate | The day of the endoscopic procedure
  This is defined as the absence of residual visible tissue after endoscopic resection
En-bloc endoscopic resection rate | The day of the endoscopic procedure
  This is defined as a single piece endoscopic resection, with clear margins
Incidence of procedure-related technical complications (Safety of the technique) | The day of the endoscopic procedure
  This will be defined as any complication occuring during the performance of the endoscopic procedure, such as muscle galling, rectal muscle perforation, minor or major bleeding, anesthesia-related adverse events, endoscopic material defect
Incidence of early procedure-related adverse events | Starting the next day following the endoscopic procedure until 30 days after the procedure
  This will be assessed by evaluating the incidence of procedure-related adverse events (AEs) and serious adverse events (SAEs) within 30 days post-procedure. This includes bleeding rates, perforation rates, infection rates among other complications.
Incidence of late procedure-related adverse events (Long-term safety of the procedure) | From the endoscopic procedure date until 5 years after the procedure date
  This will be assessed by evaluating the incidence of late procedure-related complications within 1, 3 and 5 years after the procedure. This includes delayed haemorrhage, delayed perforation, stenosis, stricture, infection and local pain among other complications
Endoscopic tumor characteristics | From the endoscopic procedure date until 5 years after the procedure date
  This will be assessed by the correlation between endoscopic tumor characteristics and the rates of recurrence and salvage surgery. Endoscopic tumor characteristics include the presence of a non-lifting sign, muscle retraction sign, fibrosis, and the description of vessels density (low/moderate/high)
Pathologic tumor characteristics | From the endoscopic procedure date until 5 years after the completion of the neoadjuvant therapy
  This will be assessed by the correlation between residual tumor characteristics (e.g. resected specimen surface, the presence of residual tumor, tumor differentiation, margin status, lymphovascular invasion (LVI), perineural invasion (PNI), fibrosis degree, tumor budding) and the rates of recurrence and salvage surgery
Pathological response | From the endoscopic procedure date until 5 years after the completion of the neoadjuvant therapy
  This will be assessed by the correlation between the degree of pathological response (e.g., complete, partial, or poor response) and the rates of recurrence and salvage surgery
Molecular biomarkers | From the pathologic report date until 5 years after the endoscopic procedure date
  This will be assessed by evaluating molecular biomarkers such as Next Generation Sequencing (NGS) on the resected specimen, and correlating these findings with the rates of recurrence and salvage surgery
Survival Outcomes | From the endoscopic procedure date until 5 years after the completion of the neoadjuvant therapy
  Overall survival (OS) and disease-free survival (DFS) at 1, 3 and 5 years.

OTHER OUTCOMES:
Procedure Duration | The day of the endoscopic procedure
  The average time taken to perform the endoscopic resection, measured in minutes and reported by the endoscopist
Length of Hospital Stay | From the endoscopic procedure date to the date of the patient's discharge from the hospital, up to 30 days
  Number of days patients are hospitalized post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Saint Pierre, Brussels, Belgium